CLINICAL TRIAL: NCT06603324
Title: Efficacy and Safety of Paediatric CVVHD Treatment With MultiFiltratePRO: A Prospective Multicenter Study
Brief Title: Analysis of Paediatric Treatments With multiFiltratePRO
Acronym: ECHOped
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Collaborators: Alcedis GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVVHD-PED-01-EU
Record Dates: First submitted 2024-02-22; First posted 2024-09-19 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Renal Failure; CVVHD
Keywords: Acute Kidney Injury; Renal Replacement Therapy; Haemodiafiltration; Contintious kidney replacement therapy; Paediatric
MeSH Terms: conditions — Renal Insufficiency; Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: Treatment of acute kidney injury paediatric patients with continuous veno-venous haemodiafiltration (CVVHD) in paediatric mode with multiFiltratePRO
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CVVHD treatment in paediatric mode with multiFiltratePRO (Experimental): Treatment of acute kidney injury paediatric patients with continuous veno-venous haemodiafiltration (CVVHD) in paediatric mode with multiFiltratePRO
  Interventions: Device: CVVHD treatment in paediatric mode with multiFiltratePRO

INTERVENTIONS:
Device: CVVHD treatment in paediatric mode with multiFiltratePRO — Treatment of acute kidney injury paediatric patients with continuous veno-venous haemodiafiltration (CVVHD) in paediatric mode with multiFiltratePRO

SUMMARY:
This clinical study evaluates the performance of the MultifiltratePro in pediatric mode for Continuous Venovenous Hemodiafiltration (CVVHD) in children. Its primary aim is to assess the efficacy of the MultifiltratePro in paediatric mode, specifically in achieving at least 80% of the prescribed effluent dose within 72 hours. Additionally, the study focuses on the safety of this mode in a paediatric setting, closely monitoring for clinical adverse events, hemodynamic instability, and electrolyte imbalances. Paediatric patients with body weights between 8kg and 40kg will be treated with the MultifiltratePro for a period of up to 10 days, with the treatment duration and approach being tailored to the severity of each patient's condition.

ELIGIBILITY:
Inclusion criteria:

General:

* Paediatric Patients:
* Informed consent signed and dated by legal representative and investigator/ authorized physician.
* The minors have received the information referred to in Article 63(2) MDR in a way adapted to their age and mental maturity and from investigators or members of the investigating team who are trained or experienced in working with children.
* The explicit wish of a minor who is capable of forming an opinion and assessing the information referred to in Article 63(2) MDR to refuse participation in, or to withdraw from, the clinical investigation at any time, is respected by the investigator.

Study-specific:

* Estimated life expectancy greater than 3 days
* Children under 18 years
* Body weight ≥8kg and <40kg
* Patients with clinical indication for CVVHD

Exclusion criteria:

General:

* Any conditions which could interfere with the patient's ability to comply with the study
* Patient or legal representative is not able to give informed consent according to European Medical Device Regulation and corresponding national regulations
* In case of female patients: pregnancy or lactation period
* Participation in an interventional clinical study during the preceding 30 days
* Previous participation in the same study

Study-specific:

* Hypersensitivity to heparin or known history of heparin induced thrombocytopenia (HIT Type II)
* Uncontrolled bleeding and coagulation disorders
* Decision to limit therapeutic interventions
* Inability to establish the required vascular access

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Effluent dose | 0 hours and 72 hours after start of treatment
  Performance parameters of the paediatric treatment mode of multiFiltratePRO based on the effluent dose (prescribed vs achieved effluent dose) at 72 hours (at least 80% of the machine prescribed dose) are analysed

CONTACTS AND LOCATIONS:
Overall Officials: Michael Merker, Dr. med., Principal Investigator — Universitätsklinikum Frankfurt, Klinik für Kinder- und Jugendmedizin
Locations (1):
- Universitätsklinikum Frankfurt, Frankfurt, Germany

IPD SHARING:
Plan to Share IPD: No